CLINICAL TRIAL: NCT05548478
Title: Corneal Endothelial Cell Injury Induced by Mitomycin-C in TransEpi Single Step and Alcohol Assisted Photorefractive Keratectomy PRK: A Comparative Study
Brief Title: Corneal Endothelial Cell Injury Induced by Mitomycin-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mitomycin-C
Record Dates: First submitted 2022-09-17; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Myopia
Keywords: mytomycin
MeSH Terms: conditions — Myopia | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TransEpi single step PRK (Active Comparator)
  Interventions: Procedure: Transepithelial PRK/MMC
- alcohol assisted PRK (Active Comparator)
  Interventions: Procedure: Alcohol-Assisted PRK/MMC

INTERVENTIONS:
Procedure: Transepithelial PRK/MMC — transepithelial photorefractive keratectomy (PRK) and mitomycin C addition
  Arms: TransEpi single step PRK
Procedure: Alcohol-Assisted PRK/MMC — photorefractive keratectomy (PRK) assisted by alchol and mitomycin C addition
  Arms: alcohol assisted PRK

SUMMARY:
our study will investigate the effecacy of Mitomycin-C in TransEpi single step photorefractive keratectomy (PRK) and alcohol assisted PRK

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Primary myopia or compound myopic astigmatism.
* Preoperative manifest refraction spherical equivalent (MRSE) within the range of -1.0 to 8 D
* Stable refractive error for at least 12 months before the surgery.
* Contact lens discontinuation for at least 3 weeks.
* Estimated corneal stromal bed thickness of more than 300mm at the thinnest point

Exclusion Criteria:

* Unwilling to participate in the study.
* Previous ocular surgery
* Any diagnosed ocular disease
* History of ocular trauma

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell Density | Base line
  will be measured by Specular microscopy
Endothelial cell Density | at 1st month
  will be measured by Specular microscopy
Endothelial cell Density | at 3rd month
  will be measured by Specular microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt